CLINICAL TRIAL: NCT00098020
Title: Retinoids for Podocyte Disease
Brief Title: Podocyte Retinoids
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 050015; 05-DK-0015 (Other: NIH)
Record Dates: First submitted 2004-12-01; First posted 2004-12-02 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-10-04

CONDITIONS: Collapsing Glomerulopathy; Glomerulosclerosis, Focal Segmental
Keywords: Glomerulosclerosis; Proteinuria; Fibrosis; Chronic Kidney Disease; Nephrotic Syndrome
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental; Proteinuria; Fibrosis; Renal Insufficiency, Chronic; Nephrotic Syndrome | interventions — Isotretinoin

STUDY DESIGN:
Intervention Model Description: Phase II, open-label pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Isotretinoin (Experimental): Subjects will be treated with Isotretinoin.
  Interventions: Drug: Isotretinoin

INTERVENTIONS:
Drug: Isotretinoin

SUMMARY:
This is a pilot study of retinoids for patients with unsatisfactory response to conventional treatment of nephrotic syndrome due to focal segmental glomerulosclerosis or minimal change disease, two renal disorders associated with putatively pathogenic malfunctioning of glomerular podocytes. The hypothesis that retinoids may have reparative effects on these cells is based on previous research showing that retinoids promote the differentiation or redifferentiation of aberrant epithelial cells. Results obtained by 6 months of treatment with retinoids (that have been approved for non-renal indications) will be used as preliminary information upon which to base further testing of these agents in formal clinical trials in refractory cases of these nephrotic syndromes.

DETAILED DESCRIPTION:
Retinoids are analogues of vitamin A that regulate cellular differentiation, leading to therapeutic use in skin diseases and malignancy. In animal models of kidney diseases, retinoids restore podocyte phenotype toward normal and reduce proteinuria. The objective of this phase II trial is to evaluate safety and develop preliminary evidence of efficacy of retinoid treatment in patients with podocyte disease. The study design is an open-label trial of isotretinoin (13-cis retinoic acid). The study will be performed under the auspices of an investigational new drug (IND) from the FDA. We will enroll 10 adult patients with biopsy-proven minimal change disease (MCD), focal segmental glomerulosclerosis (FSGS), or collapsing glomerulopathy (CG). Inclusion criteria will include a prior trial of immunosuppressive therapy and proteinuria greater than or equal to 3.5 g/d while on angiotensin antagonist therapy.

The duration of the trial will be 6 months with possible additional 6-month extension for patients who only develop partial response (PR) or limited response (LR). Those who have complete response (CR) will continue the treatment for one additional month, for no more than 7 months total. Non-responders will stop at the end of 6 months. The primary clinical endpoint will be reduction in proteinuria as compared to the baseline value assessed by paired t test. The secondary clinical endpoints will be the fraction of patients who achieve CR or PR at 6 months and at one year, confirmed on urine collections four weeks apart. Retinoid therapy will be discontinued at the time a CR is confirmed, one month after the first detection of CR. Follow-up will last one year after cessation of drug therapy. Patients who have had a CR or PR but experience a relapse with >2.0g/g proteinuria during follow-up will be eligible for further retinoid therapy. Patients will undergo a renal biopsy prior to initiating therapy, in order to evaluate the extent of glomerular injury and interstitial fibrosis, unless they have had a kidney biopsy within the preceding 24 months that is available for review. Laboratory endpoints will include serum and urine cytokine levels and urine levels of podocyte proteins, including nephrin. Toxicity screening will include serum and urine chemistries, psychological profiles, radiographic films of cervical, thoracic spines and calcanei, and bone mass assessment with dual photon excitation absorptiometry (DEXA) at spine and hip.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients with podocyte diseases, MCD, FSGS (including primary, secondary, and adaptive variants), and CG (including HIV-associated variant), who meet the following criteria:

  --An adequate renal biopsy, defined as having minimum 10 glomeruli for light microscopy and minimum 3 glomeruli for electron microscopy, unless the podocyte disease is diagnostic on fewer glomeruli. Patients who have non-diagnostic or technically inadequate biopsies will be offered the opportunity to undergo a research biopsy to determine eligibility. For some patients who have had a non-diagnostic or technically inadequate biopsy, a repeat renal biopsy may be clinically indicated in an effort to diagnose and treat a potentially serious kidney disease.
* Greater than or equal to 16 years of age. The rationale for excluding younger children is that retinoids may carry greater toxicity in children, as there are reports of premature epiphyseal closure, development of slender long bones, and periostal thickening.
* Prior treatment with at least two immunosuppressive agents that have been shown to induce remission in MCD and FSGS: glucocorticoids, cyclosporine, tacrolimus, cyclophosphamide, chlorambucil, and mycophenolate mofetil. Therapy with each agent must last at least 8 weeks. Exemptions will be made for those with contraindications to these medications or those who cannot tolerate these medications. The rationale is to recruit patients who have failed conventional therapy. All patients will be off immunosuppression for at least 4 weeks before starting retinoids in order to avoid a confounding effect.
* Three first void urine protein/creatinine ratios > 2 g/g obtained within one month prior to enrolling in the study. These urine collections will be obtained after the patient has been on a stable dose of angiotensin converting enzyme(ACE) inhibitor or angiotensin receptor blocker (ARB) for at least 4 weeks (the maximal antiproteinuric effect of these medications occurs after 4 weeks). The rationale is that patients with nephrotic-range proteinuria are at high risk for progressive renal disease, justifying participation in a clinical trial with novel agents. Patients with steroid-sensitive frequently relapsing MCD will not be required to have used ACE inhibitor or ARB, as steroids alone are typically sufficient therapy to induce remission.
* If hypertensive: blood pressure of less than or equal to 140/90 on a stable dose of ACE inhibitor or ARB for at least 1 month or greater than or equal to 75 percent of measurements before the entry of the study. The rationale is that uncontrolled hypertension can exacerbate proteinuria.

EXCLUSION CRITERIA:

* Pregnancy, breastfeeding, or unwillingness to use at least two contraceptive methods (at least one of which must be primary, including tubal ligation, partner vasectomy, oral contraceptives, implanted contraceptives, and intrauterine device). The rationale is that retinoids are teratogenic and are excreted in breast milk.
* Abnormal liver function test, including aspartate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin, or protime. The rationale is that retinoids can be hepatotoxic. The only exception will be the following: if the cause of abnormality of liver function tests (LFT) is felt to be due to a specific hepatotoxic drug such as a statin and the levels are less than 2 times the upper limit of the normal AND normalize upon holding the offending drug, patients may be considered for study participation after consultation with hepatology service.
* Hypertriglyceridemia greater than 500 mg/dL despite statin/fibrate therapy. The rationale is that retinoids can increase lipids, particularly triglyceride as this can lead to pancreatitis.
* Any medical conditions requiring concurrent immunosuppression, as this pilot study is designed to evaluate the effect of retinoids as a monotherapy.
* Any medical conditions requiring concurrent use of tetracycline, minocycline, or doxycycline, due to enhanced risk of increased intracranial pressure.
* Hypersensitivity to retinoids.
* Presence of any unstable cardiovascular disease, uncontrolled diabetes with hemoglobin A1c greater than 8 percent, chronic inflammatory or infectious conditions except HIV-1 infection. Retinoids have been associated with chest pain of unclear etiology, increased serum glucose, myelosuppression and increased risk of infection. The etiology of infection is not clear but may be related to myelosuppression.
* Those with HIV-1 infection must not have any evidence for opportunistic infectious complications and have cluster of differentiation 4 (CD4) count greater than or equal to 200. Both tretinoin and isotretinoin have been safely studied in HIV-infected patients for other indications.
* glomerular filtration rate (GFR) less than 40 ml/min/1.73m(2) estimated by 5-variable Modification of Diet in Renal Disease (MDRD) equation, as the metabolites of retinoids are excreted in part in urine, and there is a concern for increased toxicity. In participants less than 18 years of age, we will use Schwartz equation.
* Expansion of glomerulus or interstitial formation on the biopsy.
* Untreated depression, as retinoids have been associated with depression, suicidal ideation, and aggressive behavior. If patients manifest significant depressive symptoms, they will be included in the study only if assessed and agreed by a psychiatrist (either at NIH or other) and if they have regular follow-up visits with a psychiatrist.
* Factors that increase the risk of renal biopsy. These include the following: unwillingness to accept blood transfusion, bleeding diathesis, single kidney, small kidneys (less than 9.5 cm).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2004-11-26; Primary Completion 2016-06-27 (Actual); Study Completion 2016-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey B Kopp, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
The stored samples for this trial include plasma, urine, and renal biopsy samples. The plasma and urine are collected for cytokine measurement. Renal biopsy is done to evaluate histologic and ultrastructural changes. Samples/Data will be shared with collaborating investigators.
Time Frame: Until study closure.
Access Criteria: Collaborating investigators

REFERENCES:
- [Background] WILSON JG, ROTH CB, WARKANY J. An analysis of the syndrome of malformations induced by maternal vitamin A deficiency. Effects of restoration of vitamin A at various times during gestation. Am J Anat. 1953 Mar;92(2):189-217. doi: 10.1002/aja.1000920202. No abstract available. PMID 13030424
- [Background] Lelievre-Pegorier M, Vilar J, Ferrier ML, Moreau E, Freund N, Gilbert T, Merlet-Benichou C. Mild vitamin A deficiency leads to inborn nephron deficit in the rat. Kidney Int. 1998 Nov;54(5):1455-62. doi: 10.1046/j.1523-1755.1998.00151.x. PMID 9844121
- [Background] Kriz W, Elger M, Nagata M, Kretzler M, Uiker S, Koeppen-Hageman I, Tenschert S, Lemley KV. The role of podocytes in the development of glomerular sclerosis. Kidney Int Suppl. 1994 Feb;45:S64-72. No abstract available. PMID 8158902
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2005-DK-0015.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Isotretinoin: Subjects will be treated with isotretinoin initially at 1mg/kg for the first 4 weeks and then dose will escalate to a higher dose only if subjects have tolerated the lower dose.
  In younger patients of 16 and 17 years of age, the dose will be started at 1 mg/kg and will remain at this dose without escalation.
Period: Overall Study
Arm/Group | Isotretinoin
Started | 12
Started Isotretinoin | 8
Completed | 6
Not Completed | 6
Not completed — Adverse Event | 2
Not completed — Lost to Follow-up | 1
Not completed — elevated liver enzymes | 1
Not completed — Low urine PCR | 1
Not completed — Low epidermal growth factor receptor | 1

BASELINE CHARACTERISTICS:
Groups:
- Isotretinoin: subjects will be treated with iIsotretinoin.
Arm/Group | Isotretinoin
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 9
  More than one race | 0
  Unknown or Not Reported | 1
Protein, Urine [Mean (Standard Deviation); unit: mg/dL] | 626.42 (642.58)
Creatinine, Urine [Mean (Standard Deviation); unit: mg/dL] | 71.37 (43.36)
Protein/Creatinine Ratio, Urine [Mean (Standard Deviation); unit: g/g] | 8.42 (4.69)

OUTCOME MEASURES:

1. Primary Outcome: Change in Proteinuria at Week 24 From Baseline
Description: Change of proteinuria at Week 24 compared to the baseline using protein/creatinine ratio (PCR)
Time Frame: Baseline and Week 24
Population: A total of 7 patients is analyzed due to 1 withdrawal.
Measure: Mean (Standard Deviation); unit: g/g
Groups:
- Isotretinoin: oral isotretinoin
Arm/Group | Isotretinoin
Number analyzed (Participants) | 7
g/g
  Baseline | 8.42 (4.69)
  Week 24 | 7.67 (5.36)

2. Secondary Outcome: Number of Patients Who Are in Complete Remission (CR) or Partial Remission (PR) at 6 Months or at the End of One Year.
Description: Based on 24hour proteinuria, response outcomes are defined as CR (complete remission): <0.3 g/g PR (partial remission): 50% fall from baseline and <2.0 g/g
Time Frame: End of one year from baseline
Population: Seven out of 8 subjects who were treated with isotretinoin completed Week 24. One out of the 7 subjected who completed Week 24 did not complete the whole study.
Measure: Count of Participants; unit: Participants
Arm/Group | Isotretinoin
Number analyzed (Participants) | 7
Participants | 0

ADVERSE EVENTS:
Time Frame: 18 months
Groups:
- Isotretinoin: Subjects will be treated with isotretinoin .
Arm/Group | Isotretinoin
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Isotretinoin (N=8)
Agitation (Nervous system disorders) | 1 (3)
Alanine aminotransferase increased (Renal and urinary disorders) | 1 (1)
Alopecia (Blood and lymphatic system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (3)
Anorexia (Gastrointestinal disorders) | 2 (2)
Arthralgia (knee/ankle) (Immune system disorders) | 1 (1)
Ascites (Blood and lymphatic system disorders) | 1 (1)
Aspartate aminotransferase increased (Hepatobiliary disorders) | 1 (1)
Cholesterol high (Hepatobiliary disorders) | 1 (1)
Conduction disorder (General disorders) | 1 (1)
Creatinine Increased CTCAE (Renal and urinary disorders) | 1 (1)
Creatinine increased (Renal and urinary disorders) | 1 (2)
Dexamethasone x4 doses: start MMF and CSA (General disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2)
Dry skin (lips) (Skin and subcutaneous tissue disorders) | 2 (4)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Edema Limbs (Blood and lymphatic system disorders) | 3 (4)
Edema Trunk (Blood and lymphatic system disorders) | 1 (1)
Epistaxis (Blood and lymphatic system disorders) | 1 (1)
Facial pain (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 4 (4)
Headache (General disorders) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (2)
Hoarseness (General disorders) | 1 (1)
Hyperkalemia (Renal and urinary disorders) | 2 (6)
Hypertension (Cardiac disorders) | 3 (3)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Night Blindness (Eye disorders) | 1 (1)
Pacemaker placed (Cardiac disorders) | 1 (1)
Periorbital edema (Blood and lymphatic system disorders) | 1 (2)
Postnasal drip (Infections and infestations) | 1 (1)
Productive cough (Infections and infestations) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Scalp pain (General disorders) | 2 (2)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Vasovagal reaction (Cardiac disorders) | 1 (1)
Watering eyes (General disorders) | 1 (1)
Weight loss (Metabolism and nutrition disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes